CLINICAL TRIAL: NCT04745780
Title: Randomized, Controlled, Open-label Study to Evaluate the Efficacy and Safety of a Combination Containing Myo-inositol, D-chiro-inositol, Alpha-lactalbumin, Zinc and Extract of Gymnema Sylvestre in Subjects With Type 2 Mellitus Diabetes.
Brief Title: Evaluation of Efficacy and Safety of a Combination Containing Myo-inositol, D-chiro-inositol, Alpha-lactalbumin, Zinc and Extract of Gymnema Sylvestre in Subjects Diabetic Patients.
Acronym: MYDIAGYM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MYO_DCI_GYM_DIABETES
Record Dates: First submitted 2021-02-05; First posted 2021-02-09 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Myo-inositol; Gymnema sylvestre
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Inositol; Zinc; Lactalbumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Arm (Experimental): Treated with a formulation containing Myo-inositol (1950 mg), D-chiro-inositol (50 mg), Gymnema sylvestre (250 mg), Zinc (7,5 mg) and Alpha-lactalbumin (50 mg) - Two-times daily on an empty stomach, for 6 months.
  Interventions: Dietary Supplement: Myo-inositol, D-chiro-inositol, Gymnema sylvestre, Zinc and Alpha-lactalbumin
- Placebo Arm (Placebo Comparator): Treated with Placebo - Two-times daily on an empty stomach, for 6 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Myo-inositol, D-chiro-inositol, Gymnema sylvestre, Zinc and Alpha-lactalbumin — Myo-inositol (1950 mg), D-chiro-inositol (50 mg), Gymnema sylvestre (250 mg), Zinc (7,5 mg) and Alpha-lactalbumin (50 mg) - Two-times daily on an empty stomach, for 6 months
  Arms: Study Arm
Dietary Supplement: Placebo — Placebo - Two-times daily on an empty stomach, for 6 months
  Arms: Placebo Arm

SUMMARY:
Mellitus type 2 diabetes (T2MD) is a chronic disease characterized by high glucose plasmatic level due to an alteration of insulin function. Several authors have correlated this altered function to an inositol depletion. The main present member of inositol family in biological systems is undoubtedly myo-inositol, a precursor of several second messengers, widely involved in insulin signalling. For this reason this molecule is considered an insulin-sensitizer. The high excretion of inositol in T2MD patients is frequent, inducing a myo-inositol depleted state that favours the onset of insulin resistance, impairing the activity of this hormone. The aim of this study is to evaluate the efficacy and the safety of a food supplement containing myo-inositol in T2MD patients.

ELIGIBILITY:
Inclusion Criteria:

* With diagnosis of Type 2 Mellitus Diabetes for at least 1 year
* Levels of Hb1Ac ranging from 7.5% to 9.0%

Exclusion Criteria:

* Patients that require insulin treatment
* Treated at baseline with food supplements or drugs containing Myo-inositol, D-chiro-inositol, alphalactalbumin, zinc, or Gymnema Sylvestre;
* Any contraindications to the treatment or to any substance used for the treatment
* Subjects with intestinal malabsorption
* Patients subjected to surgery within 6 months before baseline;
* Chronic treatment with systemic corticosteroids

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | up to 6 months of treatment
  Variation of glycated hemoglobin level (HbA1c) after 3 and 6 months in comparison to baseline detected in the blood - %

SECONDARY OUTCOMES:
Glycemia | At baseline and 3 and 6 months of treatment
  Variation of fasting blood sugar level after 3 and 6 months in comparison to baseline detected in the blood - mg/dL
Cholesterol | At baseline and 3 and 6 months of treatment
  Variation of cholesterol level (Total, HDL and LDL) after 3 and 6 months in comparison to baseline detected in the blood - mg/dL
Hypoglycemic events | At baseline and 3 and 6 months of treatment
  Number of hypoglycemic events (< 70 mg/dl) and severe hypoglycemic events (< 54 mg/dl) during the study (6 months) - Number of events (n)

CONTACTS AND LOCATIONS:
Locations (1):
- Basilio Pintaudi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No